CLINICAL TRIAL: NCT01397838
Title: Phase 1 Study of an Oral Pro-boneTM, Administered to Post Menopausal Osteopenic Women
Brief Title: Safety Study of an Oral Pro-boneTM, Administered to Post Menopausal Osteopenic Women
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: OsteoBuild Ltd. (Industry)
Responsible Party: Prof. Boris Kaplan, Rabin Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: OBCS-001
Record Dates: First submitted 2011-07-18; First posted 2011-07-20 (Estimated); Last update posted 2011-07-20 (Estimated); Status verified 2011-07

CONDITIONS: Osteopenia
Keywords: Osteopenia
MeSH Terms: conditions — Bone Diseases, Metabolic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pro-Bone (Experimental)
  Interventions: Drug: Pro-Bone

INTERVENTIONS:
Drug: Pro-Bone — 500 mg Capsules of Pro-Bone twice daily

SUMMARY:
Recent studies have shown that inhibition of Aquaporine-9 channels may ameliorate the bone degradation process. Pro-bone is an AQ - 9 channels inhibitor. This study is design to evaluate the safety of Pro-bone.

ELIGIBILITY:
Inclusion Criteria:

* BMD as measured by DEXA at screening, should range between (-1)to (-2.5) SD from normal values.
* At least 12 months of spontaneous amenorrhea or at least 6 weeks postsurgical bilateral oophorectomy with or without hysterectomy.
* Study participants not taking estrogen alone or estrogen/progestin containing drug products.
* Study participants not taking any anti-osteoporosis treatment for at list one year.
* The following washout periods should be before baseline assessments are made for subjects previously on estrogen alone or estrogen/progestin containing products:

  1. 8 weeks or longer for any prior use of estrogen and/or progestin products.
  2. 6 months or longer for prior progestin injectable drug therapy.
  3. Women between 45 and 65 years (inclusive) of age.
  4. BMI 22-30 (inclusive)
  5. Non-smoking (by declaration) for a period of at least 6 months.
  6. Subjects able to adhere to the visit schedule and protocol requirements and be available to complete the study.
* Subjects who provide written informed consent.

Exclusion Criteria:

* Women have documentation of a positive screening mammogram (obtained at screening or within 9 months of study enrolment) or abnormal clinical breast examination prior to enrolment in clinical studies.
* Known history of significant medical disorder, which in the investigator's judgment contraindicates administration of the study medications.
* Any clinically significant abnormality, upon physical examination or in clinical laboratory test, at screening visit.
* Known history of drug or alcohol abuse according to participant declaration at screening visit.
* Any acute medical situation (e.g. acute infection) within 48 hours of study start, which is considered of significance by the Principal Investigator.
* Subjects who are non-cooperative or unwilling to sign consent form.

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2011-09; Primary Completion 2011-12 (Estimated); Study Completion 2012-01 (Estimated)

PRIMARY OUTCOMES:
Adverse events recorded throughout the study | 4 weeks
Blood and urinalysis values assessed at pre-dose and according to study design. | 4 weeks

SECONDARY OUTCOMES:
Vital signs | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Boris Kaplan, Prof., Principal Investigator — Rabin Medical Center